CLINICAL TRIAL: NCT00997893
Title: Effects of Estradiol and Soy on Menopausal Symptoms
Brief Title: Research Investigation of Soy and Estrogen
Acronym: RISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Pauline M. Maki, Ph.D, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-0052; 5R01MH083782-05 (NIH)
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Results first posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Menopause; Hot Flashes
Keywords: menopause; hot flashes; soy; estrogen; anxiety
MeSH Terms: conditions — Hot Flashes; Anxiety Disorders | interventions — Estradiol; Estrogens; Medroxyprogesterone Acetate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Estradiol/Medroxyprogesterone Acetate (Experimental): 1 mg/d oral Estradiol pill and 0 mg/d oral placebo pill for 12 weeks, followed by 10 mg/d oral medroxyprogesterone acetate (MPA) pill, for 10 days.
  Interventions: Drug: Estradiol; Drug: Medroxyprogesterone Acetate (MPA); Drug: Soy Placebo
- Soy Phytoestrogen (Experimental): 55 mg/twice daily oral Novasoy®/Soy Phytoestrogen pill for 12 weeks, followed by 0 mg/d oral placebo pill, for 10 days.
  Interventions: Dietary Supplement: Soy Phytoestrogen; Drug: MPA Placebo
- Placebo (Placebo Comparator): 0 mg tablet/twice daily oral placebo pill for 12 weeks, followed by 0 mg/d oral placebo pill, for 10 days.
  Interventions: Drug: Soy Placebo; Drug: MPA Placebo

INTERVENTIONS:
Dietary Supplement: Soy Phytoestrogen — Novasoy® pill (55 mg)
  Other Names: NovaSoy 400
  Arms: Soy Phytoestrogen
Drug: Estradiol — Estradiol pill (1 mg)
  Other Names: estrogen, estradiol acetate
  Arms: Estradiol/Medroxyprogesterone Acetate
Drug: Medroxyprogesterone Acetate (MPA) — medroxyprogesterone acetate (MPA) (10mg)
  Other Names: MPA
  Arms: Estradiol/Medroxyprogesterone Acetate
Drug: Soy Placebo — oral placebo pill (0mg Soy Phytoestrogen)
  Other Names: sugar pill
  Arms: Estradiol/Medroxyprogesterone Acetate; Placebo
Drug: MPA Placebo — oral placebo pill (0mg MPA)
  Other Names: sugar pill
  Arms: Placebo; Soy Phytoestrogen

SUMMARY:
The purpose of this study is to determine the effects of oral estradiol and soy phytoestrogens on anxiety, stress responsivity and cognition in perimenopausal women.

DETAILED DESCRIPTION:
Anxiety is a common, but understudied complaint in midlife women, and increases during the menopausal transition. Changes in estrogen are dramatic during the menopausal transition, and indirect data suggest a potential role for estrogen, particularly estrogen receptor beta, in mediating anxiety. Two subtypes of the estrogen receptor, alpha and beta (ER-alpha and ER-beta), appear to be critically involved in the expression of anxiety in females. Compounds that preferentially target ER-beta, including plant-derived estrogens (phytoestrogens), lower both anxiety behaviors and responsivity to discrete stressors, including social stress, in laboratory animals. The primary aim of this proposal is to carry out the first study to translate these preclinical studies to humans by comparing and contrasting of the effects of phytoestrogens, estradiol, and placebo on daily anxiety and responses to moderate psychosocial stress in the laboratory. As second focus is emotional and non-emotional cognition. This focus stems from evidence that estrogen can protect against the negative impact of glucocorticoids on memory. These aims will be accomplished in a 12-week randomized placebo-controlled, clinical trial comparing three treatments: 1) a phytoestrogen supplement (Novasoy® 400, 55 mg tablet twice daily); 2) oral estradiol (1 mg/daily; plus 10 mg medroxyprogesterone acetate at study end 10 for 10 days); and 3) placebo (identical appearing tablets twice daily). The enrollment target is 120 healthy women in the menopausal transition (40 per group). To measure anxiety, women will complete the State-Trait Anxiety Inventory (STAI). To measure responsivity to psychosocial stress, parallel forms of the Trier Social Stress Test, a widely used laboratory induction that involves unanticipated public speaking and social evaluative fear, will be used to induce moderate psychosocial stress before and after treatment. At both laboratory sessions, measures of subjective stress (STAI), cortisol, and emotional memory performance will be obtained at multiple points during a control condition and during the psychosocial stress condition. Lastly, we will measure treatment effects on measures of verbal memory.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Perimenopausal as defined by the Stages of Reproductive Aging Workshop (STRAW) criteria, specifically in either of the two following stages: a) early transition defined as changes in cycle length of seven days or more in either direction in consecutive cycles or b) late transition defined as > 60 days amenorrhea and FSH > 40 IU/mL
* Intact uterus/ovaries (i.e. no surgical menopause)
* at least 1 self-reported hot flash per week
* Estrogen therapy not contraindicated
* Able to give informed consent
* Age between 40 and 65 years
* English as first and primary language

Exclusion Criteria:

* Positive pregnancy test or breastfeeding (pregnancy tests will be given to all women)
* Obesity > 35 BMI
* Previous history of endometrial hyperplasia/neoplasia
* Previous history of cancers of the breast or reproductive tract
* History of presence of myocardial infarction (MI) or stroke
* Current clinical diagnosis or a diagnosis within the past year of an anxiety disorder, severe recurrent depression, or severe psychiatric disturbance
* History of head injury with more than 60 minutes loss of consciousness
* History of neurological condition affecting cognitive function (e.g., brain tumor, multiple sclerosis)
* History of developmental disability affecting cognitive function (e.g., mental retardation, attention deficit)
* Current use of CNS-acting medication (e.g., antidepressants, anxiolytics, diphenhydramine)
* History or presence of cerebrovascular accident, sickle cell anemia
* History of alcohol or drug abuse as defined by DSM criteria
* Abnormal vaginal bleeding of undetermined cause
* Untreated or uncontrolled hypertension defined as systolic blood pressure greater than 165 mm hg or diastolic blood pressure greater than 95 mm hg
* Concurrent administration of medication containing estrogen, progestin, SERM within four months of enrollment
* Concurrent administration of medication containing St. John's wort, bisphosphonates, or dietary phytoestrogens within one month of enrollment
* History of migraine associated with hormone use
* History or presence of deep vein thrombosis, thrombophlebitis or thromboembolic disorder
* Current participation in any other clinical trial within 30 days of enrollment
* Smoker
* Diabetes
* Premature ovarian failure (defined as having last menstrual period before age 40)
* Abnormal PAP smear in previous year
* Abnormal mammogram in previous year
* Vegans (vegetarians who tend to consume greater than average doses of phytoestrogens)
* Allergy to soy (affects ~1% of people in the United States; reactions are typically mild)
* Symptomatic fibroids (significant size or significant menstrual changes)
* Menorrhagia
* Lactose intolerant

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pauline M Maki, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UIC Department of Psychiatry Women's Mental Health Research Program Website — https://www.psych.uic.edu/research/womens-mental-health-research-program

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 63 of the 96 enrolled subjects met the post-enrollment eligibility criteria. Twenty-three of 63 enrolled subjects withdrew prior to randomization. A total of 40 subjects were randomized.
Period: Overall Study
Arm/Group | Estradiol/Medroxyprogesterone Acetate | Soy Phytoestrogen | Placebo
Started | 14 | 13 | 13
Completed | 12 | 12 | 13
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Unable to meet study timelines | 1 | 0 | 0
Not completed — Pain/pain meds during Visit 4 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Estradiol/Medroxyprogesterone Acetate: 1 mg oral estradiol for 12 weeks followed by 10 mg/d oral MPA
- Phytoestrogen: 55 mg Novasoy pill b.i.d. (Total daily dose 110 mg)
- Placebo: Placebo pill b.i.d. (0 mg Novasoy® and 0 mg estradiol)
- Total: Total of all reporting groups
Arm/Group | Estradiol/Medroxyprogesterone Acetate | Phytoestrogen | Placebo | Total
Number analyzed (Participants) | 14 | 13 | 13 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 13 | 40
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.07 (4.16) | 51.38 (3.90) | 49.31 (3.84) | 50.25 (3.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 13 | 40
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 13 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in STAI-6 Score
Description: STAI-6; State-Trait Anxiety Inventory- Short Form is a measure of anxiety where higher scores indicate higher/elevated anxiety. Minimum value 6 is and maximum value is 24.
Time Frame: Week 0, 10, 12, and 16-18
Measure: Mean (Standard Error); unit: score on STAI scale
Groups:
- Phytoestrogen: 55 mg Novasoy pill b.i.d.
- Placebo: Placebo pill b.i.d
Arm/Group | Estradiol/Medroxyprogesterone Acetate | Phytoestrogen | Placebo
Number analyzed (Participants) | 14 | 13 | 13
score on STAI scale
  Baseline (Week 0) | 12.31 (0.74) | 11.85 (0.74) | 10.76 (0.76)
  Early-Treatment(Week 10) | 11.69 (0.73) | 11.38 (0.71) | 11.24 (0.74)
  Late-Treatment(Week 12) | 12.88 (0.75) | 10.99 (0.72) | 10.55 (0.75)
  Post-Treatment (Week 16-18) | 11.84 (0.74) | 11.19 (0.72) | 11.15 (0.76)
Statistical Analysis 1: Comparison: Estradiol/Medroxyprogesterone Acetate vs Phytoestrogen vs Placebo; Test type: Other; p = .004, Mixed Models Analysis — treatment x time p=.004; A mixed effects regression model (Estimation method=maximum likelihood; Random intercept) was conducted to compare the effects of phytoestrogens and estradiol to placebo. Primary predictor variables in the model included treatment and time, as well the treatment by time interaction

2. Primary Outcome: Changes in STAI-6 Scores Before and After Psychosocial Stressor Over Time
Description: as for outcome 1
Time Frame: Baseline (Week 0) and Treatment (Week 12)
Measure: Mean (Standard Error); unit: score on STAI scale
Arm/Group | Estradiol/Medroxyprogesterone Acetate | Phytoestrogen | Placebo
Number analyzed (Participants) | 14 | 13 | 13
score on STAI scale
  Baseline (Week 0), Before Stressor | 8.73 (0.89) | 8.69 (0.89) | 9.77 (0.89)
  Baseline (Week 0), After Stressor | 12.61 (0.89) | 12.92 (0.89) | 12.23 (0.89)
  Post-Treatment (Week 12), Before Stressor | 8.25 (0.94) | 10.87 (0.91) | 9.61 (0.89)
  Post-Treatment (Week 12), After Stressor | 13.70 (0.94) | 15.37 (0.91) | 12.69 (0.89)
Statistical Analysis 1: Comparison: Estradiol/Medroxyprogesterone Acetate vs Phytoestrogen vs Placebo; Test type: Other; p = .98, Mixed Models Analysis — visit x time x treatment interaction p=.98; A mixed effects regression model (Estimation method=maximum likelihood; Random intercept) was conducted to compare the effects of phytoestrogens and estradiol to placebo before and after a psychosocial stressor. Predictor variables in the model included treatment, time (before and after the psychosocial stressor), visit (Baseline, 12 weeks), and all two and three way interactions

3. Primary Outcome: Memory for Emotionally Valent Words and Neutral Words
Description: Proportion correct out of 18 word pairs (6 positive, 6 negative and 6 neutral) after laboratory-induced stress using Trier Social Stress Test (TSST). Maximum score is 18 and minimum score is 0; higher scores indicate a better score.
Time Frame: Baseline (Week 0) and Treatment (Week 12)
Measure: Mean (Standard Error); unit: Proportion Correct
Arm/Group | Estradiol/Medroxyprogesterone Acetate | Phytoestrogen | Placebo
Number analyzed (Participants) | 14 | 13 | 13
Proportion Correct
  Baseline (Week 0)- Control | 0.45 (0.08) | 0.45 (0.08) | 0.38 (0.08)
  Baseline (Week 0)- TSST | 0.48 (0.08) | 0.40 (0.08) | 0.47 (0.08)
  Post-Treatment (Week 12)- Control | 0.47 (0.08) | 0.42 (0.08) | 0.37 (0.08)
  Post-Treatment (Week 12)-TSST | 0.51 (0.08) | 0.46 (0.08) | 0.44 (0.08)
Statistical Analysis 1: Comparison: Estradiol/Medroxyprogesterone Acetate vs Phytoestrogen vs Placebo; Test type: Other; p = .68, Mixed Models Analysis — treatment x time (before and after the psychosocial stressor) x visit p=.68; A mixed effects regression model (Estimation method=maximum likelihood; Random intercept) was conducted to compare the effects of phytoestrogens and estradiol to placebo on emotional memory following a laboratory induced stress. Primary predictor variables in the model included treatment, time (before and after the psychosocial stressor), visit (Baseline, 12 weeks), and all two and three way interactions

4. Primary Outcome: Change in Verbal Memory, Immediate Recall
Description: Immediate recall on the Logical Memory subset of the Wechsler Memory Scale-Revised, in which higher scores indicate a better recall and outcome. The minimum value is 0 and maximum value is 25.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: test scores on the Logical Memory test
Arm/Group | Estradiol/Medroxyprogesterone Acetate | Phytoestrogen | Placebo
Number analyzed (Participants) | 14 | 13 | 13
test scores on the Logical Memory test | -.02 (0.87) | 2.31 (0.82) | 2.08 (0.82)
Statistical Analysis 1: Comparison: Estradiol/Medroxyprogesterone Acetate vs Phytoestrogen vs Placebo; Test type: Other; p = .11, Mixed Models Analysis — treatment x time p=.11; A mixed effects regression model (Estimation method=maximum likelihood; Random intercept) was conducted to compare the effects of phytoestrogens and estradiol to placebo on verbal memory (logical memory; immediate). Primary predictor variables in the model included treatment and time, as well the treatment by time interaction

5. Primary Outcome: Change in Verbal Memory, Delayed Recall
Description: Delayed recall on the Logical Memory subset of the Wechsler Memory Scale-Revised, in which higher scores indicate a better recall and outcome. The minimum value is 0 and maximum value is 25.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: Test scores on the Logical Memory test
Arm/Group | Estradiol/Medroxyprogesterone Acetate | Phytoestrogen | Placebo
Number analyzed (Participants) | 14 | 13 | 13
Test scores on the Logical Memory test | .87 (1.03) | 1.61 (0.96) | 1.08 (0.96)
Statistical Analysis 1: Comparison: Estradiol/Medroxyprogesterone Acetate vs Phytoestrogen vs Placebo; Test type: Other; p = .86, Mixed Models Analysis — treatment x time p=.86; A mixed effects regression model (Estimation method=maximum likelihood; Random intercept) was conducted to compare the effects of phytoestrogens and estradiol to placebo on verbal memory (logical memory; immediate)Primary predictor variables in the model included treatment and time, as well the treatment by time interaction

ADVERSE EVENTS:
Time Frame: Adverse event reporting forms have been completed for all participants reporting adverse events during bi-weekly phone safety screenings (Week 2, 4, 6 and 8), as well as in person visits during Week 10, and Week 12.
Arm/Group | Estradiol/Medroxyprogesterone Acetate | Phytoestrogen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/14 | 0/13 | 0/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol/Medroxyprogesterone Acetate (N=14) | Phytoestrogen (N=13) | Placebo (N=13)
Non-serious; irregular uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) — Participant had heavy and moderate uterine bleeding. Exam and transvaginal ultrasound was performed. Possible hyperplasia was found and later biopsied with benign results. Event was self reported by participant.

LIMITATIONS AND CAVEATS:
Enrollment goals of 120 women were not met. Many declined to participate due to concerns about the safety of taking estrogens (the study was performed shortly after publication of the Women's Health Initiative) and due to the time commitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No